CLINICAL TRIAL: NCT02789735
Title: Effectiveness of Low Level Laser Therapy in Persistent Pregnancy-related Pelvic Girdle Pain After Childbirth
Brief Title: Low Level Laser Therapy in Persistent Pelvic Girdle Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LLLT
Record Dates: First submitted 2016-04-08; First posted 2016-06-03 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Pelvic Girdle Pain
Keywords: Pregnancy; laser therapy; persistent pain; pelvic pain
MeSH Terms: conditions — Pelvic Girdle Pain; Pelvic Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device: LiteCure LCT-1000® (Active Comparator): Treatment with 10 J/cm²
  Interventions: Device: Active laser therapy
- Device: Sham LiteCure (Sham Comparator): Sham i.e. visible red light
  Interventions: Device: Sham laser therapy

INTERVENTIONS:
Device: Active laser therapy — Laser therapy at predetermined sites
  Other Names: Low level laser therapy
  Arms: Device: LiteCure LCT-1000®
Device: Sham laser therapy — Sham therapy at predetermined sites
  Arms: Device: Sham LiteCure

SUMMARY:
Persistent pregnancy-related pelvic girdle pain is common, 2-5% av all women given birth is suffering from disabling daily pain with high impact on quality of life.

A prospective double-blinded randomised controlled trial will be performed with a baseline assessment 7-10 months after childbirth with follow-up directly and 6 months after a treatment period with low level laser therapy (LLLT) or sham laser treatment, given at 12 planned treatment sessions during four weeks. 60 women will be included in the study.

If LLLT can reduce pain and improve function there will be a new treatment option for this condition.

DETAILED DESCRIPTION:
A prospective double-blinded randomised controlled trial will be performed with a baseline assessment 7-10 months after childbirth with follow-up directly and 6 months after a treatment period with low level laser therapy (LLLT) or sham laser treatment, given at 12 planned treatment sessions during four weeks.

A total of 60 women will be sampled consecutively. Women eligible to participate will be those women who were registered at a maternal health care unit in the municipalities of Sundsvall and Timrå with subsequent childbirth registered at the Sundsvall-Härnösand County Hospital, Sweden. An invitation letter with a prepaid response envelope will be sent by postal mail to the eligible women by contact information retrieved from the labour ward. Women who respond will be enrolled and approve their participation by signed informed consent. The women will be included in the study according to inclusion and exclusion criteria following a baseline assessment that comprises a urinary test, questionnaires and clinical examination. After inclusion a blood sample, for serum and plasma, will be drawn at inclusion and directly after the treatment period.

Randomisation and blinding The randomisation sequence will be generated by a statistician not involved in the study. Randomisation will be done using block randomisation (block size 4 or 6) without stratification. The investigators will use sequentially numbered, opaque, sealed envelopes which have been pre-prepared in advance by the statistician. Women who fulfil the inclusion criteria will be randomised to active laser treatment or sham laser treatment. A research assistant not involved in the inclusion assessments will perform the randomisation, prepare and handle the allocated treatment device before and after each treatment session. The treatment will be given by a physiotherapist who is blinded to treatment group, the women's case history, questionnaires and clinical examinations.

All collected data will be handled, stored and analysed at the Department of Public Health and Caring Sciences at Uppsala University. The analysts will be blinded to the treatment allocation until data of primary outcomes have been analysed and conclusions have been drawn and signed in writing before the code is broken.

Questionnaires At baseline, the women will complete questionnaires which include questions on socio-demographic data, somatic and mental health, gynaecological and obstetric history, and lifestyle.

At baseline and follow-ups, the women will report present pain distribution on a pain drawing (including onset and modality of pain). Pain intensity at present and as worst during the past week will be measured by a 100 mm VAS (Visual analogue scale). Functioning will be assessed by Disability Rating Index (DRI), Pelvic Girdle Questionnaire (PGQ) and Short Form 36 (SF-36). Throughout the treatment period, the women will daily record pain intensity in a pain diary by use of a 100 mm VAS.

At the follow-up after the treatment period the women will complete a Global Perceived Effect scale, report any adverse event, and report their opinion on whether or not they have received active treatment.

Clinical examination The two assessors, a gynaecologist and a physiotherapist, will perform the examinations without knowledge of assigned treatment, the women's case history, questionnaire replies and clinical examinations. The test procedure and test sequence will be the same throughout the study.

A gynaecologic examination, including an ultrasound examination, will be performed by a gynaecologist at baseline. Provoked pain by a gentle pressure on the following 13 predetermined intra-pelvic anatomical landmarks will be assessed via vaginal palpation: the coccyx, the lateral part of sacrum at the insertion of the sacrospinous ligament, the middle part of the sacrospinous ligament, the insertion of the sacrospinous ligament at the ischiadic spine, the ischium inferior to the ilio-ischial fusion and the lateral and medial part of the pubic bone. All the structures will be examined bilaterally except for the coccyx.

The musculoskeletal examinations at baseline and follow-ups will be performed by a physiotherapist. It will include examination of the lower back spine, pelvis and assessment of physical functioning. Briefly, the lower back spine will be examined by palpation of ligaments and paravertebral muscles, Kemp's foramina test, Valsalva test, SLR (straight leg raising test) and test of tendon reflexes and sensibility. The pelvis will be examined by the following tests: P4 test, Menell's test, Patrick's faber test, modified Trendelenburg test and the pubic symphysis palpation test.

Pain provocation tests will be considered positive if they duplicate or aggravate pain from the sacral area on the tested side, otherwise negative. The women will grade the provoked pain on a 100 mm VAS scale.

Physical functioning will be assessed at baseline and follow-up by the Six Minute Walk Test (6MWT), the Timed Up and Go Test (TUGT), the Active Straight Leg Raising Test (ASLR) and isometric trunk muscle tests.

Urine and blood sampling A urinary test will be sampled for test of hCG, human Chorionic Gonadotropin (pregnancy), at time of inclusion. A blood sample, for serum and plasma, will be drawn at inclusion and directly after the treatment period. The blood samples will be analysed directly for estrogen, progesterone, testosterone, sexual binding globulin, thyroid stimulating hormone and prolactin and thereafter discarded.

Treatment regimen The treatment comprises 12 treatment sessions distributed as one treatment daily at three consecutive days during the first treatment week and then three times a week every other weekday during the next three weeks. The treatment will be given by a licensed physiotherapist blinded for the allocated treatment. The treatment will start immediately after a menstrual period or within one week's time among women with regained menstrual periods, otherwise at any time convenient.

Throughout the treatment period the women will be asked to avoid pain provoking activities, the use of corticosteroid treatment, and sexual intercourse without use of safe contraception. Before each treatment the women will sign a form stating no unprotected intercourse since last treatment session. The women report use of pain medication and physical activity at the end of the treatment period.

Treatment equipment and performance A class IV low level laser (LiteCure LCT-1000®) and a similar sham laser will be used. Both devices are delivered by LiteCure, LLC, Newark, DE, USA. The active device delivers its energy by two wavelengths, 20% of the beam with 810 nm (nanometer) and 80% of the beam with 980 nm. Energy given will be tested before the start of the study and once every month, using Thor labs power meter PM100D and the photo sensor S 121 C, to make sure the device works correctly. There is also a red aiming beam with a wavelength of 650 nm and a power of 5 mW (milliwatt). The sham laser delivers solely the aiming beam.

The treatment is applied to the sacral region by a standard laser probe with a 26 mm quarts ball at the top, and to the internal pelvis by a 16 cm long fibre-containing transvaginal probe with a diameter of the bulb-shaped end of 18 mm. The physical therapist and the participant use safety eyewear during all treatment sessions and the treatment administration area is closed, have restricted access and no reflective surfaces.

During treatment at sacral points, the standard probe is moved 1 cm/second from a starting point to an end-point repeatedly during treatment time, bilaterally. The standard probe is held perpendicular to the body surface and pressed to the skin.

During treatment vaginally the physiotherapist palpates the anatomical landmarks by vaginal palpation to guide the transvaginal probe and hold it still on the treatment sites. Due to reasons of hygiene the transvaginal probe is covered by transparent plastic cover during treatment. The plastic cover is discarded and both probes are cleaned with ethanol-based surface disinfection after treatment.

Treatment locations on the outside of the pelvis The treatment on the outside of the pelvis is given on three sites defined by a given starting point and a treatment area. The starting point of treatment is described by vertical and horizontal coordinates.

Treatment locations on the inside of the pelvis

The treatment sites inside the pelvis are:

1. the sacrospinous ligament at the insertion on the ischial spine
2. at the middle of the sacrospinous ligament
3. the sacrospinous ligament at the insertion on the sacrum medially and in the level of the ischial spine

Treatment dose To deliver an appropriate dose of energy according to the best available evidence and experience, the active treatment group received LLLT with a dual wavelength of 810 nm and 980 nm and a dose of 10 J/cm² vaginally and 10 J/cm² over the sacral areas. The control group will receive sham treatment by a red aiming beam with a power of 5 mW with the same treatment time as the active treatment.

If a woman experiences a negative reaction or does not tolerate the treatment dose, the treatment will immediately be stopped. The amount of energy given at each treatment session will be recorded.

Data analysis Power calculation To show a statistically significant difference of at least 20 mm in pain intensity (considered as a clinically relevant difference) measured by visual analogue scale between the active treatment group and the control group, at least 32 women will be needed with the assumptions of type I error of 5% and type II error of 20%. To take account for data loss the investigators aim at a sample size of at least 30 women in each group, in total 60 women.

Statistical analysis The analyses of outcomes will be performed in accordance with the European Medicines Agency's Statistical Principles for Clinical Trials guidelines. Differences between the treatment groups regarding outcome measures will be analysed by regression analysis of variance on ranks. Other parametric and non-parametric statistical methods will be used whenever appropriate. Two-sided tests will be used and 5% statistical significance level will be chosen for all analyses. To provide unbiased comparisons between the groups the investigators will be perform an intention-to-treat analysis. Also, a per-protocol analysis on the women who complete the study according to the protocol will be performed.

Ethical considerations The use of the LLLT devices is approved by Swedish and European authorities (Reference number 2014/188, dated140811) and is supposed to have minimal side effects. The present study is approved by the Regional Ethical Review Board in Uppsala (Dnr 2014 / 188). All women will sign an informed consent.

To prevent potential injury or harm, the vaginal probe will be used with care. Also, a gynaecologic examination will be performed before start of study treatment. The effect of low level laser irradiation to an early pregnancy is not known; therefore potential harm will be sought minimised by a test of hCG at study inclusion. Also written statements of no sexual intercourse without safe contraception will be given before each treatment session.

The physical therapist and the participant will use safety eyewear during all treatment sessions and the treatment administration area will be closed, have restricted access and will be without reflective surfaces. Finally, our perception is that the advantages of the study treatment outweigh ethical problems. All of the researchers declare no conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

1. Ongoing sacral pain with onset during the preceding pregnancy reported on a present pain drawing
2. Pain intensity ≥40 mm as worst during the past week on a 100 mm visual analogue scale (VAS)
3. One positive pain provocation test of either Posterior Pelvic Pain Provocation (P4) test, Menell's test or Patrick's faber test
4. Provoked pain by a gentle pressure on the ischial spine, ipsilaterally to reported sacral pain, at least unilaterally

Exclusion Criteria:

1. A positive urinary human Chorionic Gonadotropin (hCG) test
2. Nerve root affection in the lumbo-sacral spine
3. Inflammatory disease with pelvic bone and/or spinal manifestation
4. Known endometriosis, gynaecologic cancer or ongoing malign disease
5. Previous surgery of the lumbar spine
6. Corticosteroid treatment during the past 6 months and during treatment
7. Incapacity to complete the questionnaires
8. Age <18 years
9. Body mass index ≥35 kg/m2
10. Intolerance to the treatment dose or negative reactions of the laser treatment
11. A new pregnancy, during treatment or between the follow-ups.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2021-02 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (100 mm VAS) Worst during the past week | Baseline to 6 months after treatment
  Change from baseline to follow-up
P4-test Pressure (1, 5, 10 or 15kg) added to provoke sacral pain | Baseline to 6 months after treatment
  Change from baseline to follow-up
6 minute walk test, 6MWT, distance (m) | Baseline to 6 months after treatment
  Change from baseline to follow-up
Disability rating index, DRI. Function past week % | Baseline to 6 months after treatment
  Change from baseline to follow-up

SECONDARY OUTCOMES:
Pain score (0-26) of provoked pain on intra-pelvic anatomical landmarks | Baseline to 6 months after treatment
  Change from baseline to follow-up
SF-36, questionnaire | Baseline to 6 months after treatment
  Change in quality of life from baseline to follow-up
Pelvic Girdle Questionnaire, PGQ, function % | Baseline to 6 months after treatment
  Change in function from baseline to follow-up
Timed Up and Go Test,TUGT, time (s) | Baseline to 6 months after treatment
  Change in seconds from baseline to follow-up
Isometric muscle tests, isometric endurance (s) | Baseline to 6 months after treatment
  Change in seconds from baseline to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Per Kristiansson, AssProf, PhD, Study Director — Uppsala University
Locations (1):
- Sundsvall Hospital, Sundsvall, Sweden

IPD SHARING:
Plan to Share IPD: No